CLINICAL TRIAL: NCT00693706
Title: Safety and Immunogenicity Study of GSK Biologicals' Cell Culture-based Influenza Virus Vaccine 1388442A Compared With US Licensed TIV in Healthy Adults
Brief Title: Safety and Immune Response Study of GSK Biologicals' Influenza Virus Vaccine 1388442A Compared With Fluarix
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 110127
Record Dates: First submitted 2008-06-02; First posted 2008-06-09 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: cell culture; Safety; Influenza; Humans; Adults; Immunogenicity; Influenza vaccine; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK 1388442A Group (Experimental): Subjects aged 18 to 49 years of age at the time of vaccination received 1 dose of GSK 1388442A vaccine at Day 0. The GSK 1388442A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Trivalent influenza vaccine GSK 138842A
- Fluarix Group (Active Comparator): Subjects aged 18 to 49 years of age at the time of vaccination received 1 dose of Fluarix® vaccine at Day 0. The Fluarix® vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix

INTERVENTIONS:
Biological: Trivalent influenza vaccine GSK 138842A — IM injection on Day 0
  Arms: GSK 1388442A Group
Biological: Fluarix — IM injection on Day 0
  Arms: Fluarix Group

SUMMARY:
The purpose of the study is to compare the safety of & immune response to a single dose of GSK Biologicals' cell-culture based influenza vaccine 138842A with that of a US licensed, egg-based trivalent influenza vaccine [Fluarix] in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* A male or non-pregnant, non-lactating female between 18 and 49 years of age at the time of vaccination
* Access to a telephone for scheduled follow-up telephone contacts
* Ability to provide written informed consent
* Healthy subjects as established by medical history and physical examination before entering into the study
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination and continue such precautions for 2 months after receipt of the study vaccine. All women will have a pregnancy test on the day of vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period
* Receipt of systemic glucocorticoids within 30 days of study enrollment
* Administration of immunosuppressant, cytotoxic, or other immune-modifying drugs (other than glucocorticoids) or irradiation within 6 months prior to study enrollment or planned administration during the study period
* Administration of immunoglobulins and/or blood products within 3 months prior to study enrollment or planned administration during the study period
* Previous vaccination against influenza (2007-2008 influenza season)
* History of anaphylactic or other allergic reaction to influenza vaccine, any other vaccine, or any vaccine component or excipient
* History of Guillain-Barre Syndrome (GBS)
* Acute disease, febrile illness, or upper respiratory infection at screening.
* History of splenectomy
* Any confirmed or suspected, acquired, congenital, or hereditary immunodeficiency or immunosuppressive condition (including human immunodeficiency virus [HIV]) based on medical history and physical examination
* Acquired or congenital coagulation disorders or known thrombocytopenia
* Current treatment with warfarin or heparin derivatives
* Known use of an analgesic or antipyretic medication within 12 hours prior to treatment for the purposes of prophylaxis of adverse events
* Any medical condition for which the US Advisory Committee on Immunization Practices recommends vaccination against influenza

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-06-02; Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Lenexa, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110127 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK 1388442A Group | Fluarix Group
Started | 101 | 99
Completed | 101 | 98
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 1388442A Group | Fluarix Group | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.1 (10.24) | 31.6 (9.77) | 32.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 106
  Male | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Solicited local symptoms were pain, redness and swelling at the injection site. Any = occurrence of a symptom regardless of intensity.
Time Frame: During the 7-day (Days 0-6) post vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the documented dose. The analysis of solicited symptoms based on the Total Vaccinated cohort included only vaccinated subjects and doses with documented safety data (i.e., symptom screen /sheet completed).
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 101 | 99
subjects
  Pain | 48 | 48
  Redness | 1 | 0
  Swelling | 1 | 0

2. Primary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Solicited general symptoms were arthralgia, fatigue, headache, muscle aches, shivering and temperature, assessed as oral temperature above or equal (≥) 38.0 degrees Celsius (°C). Any = occurrence of a symptom regardless of intensity or relationship to vaccination.
Time Frame: During the 7-day (Days 0-6) post vaccination period
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 100 | 99
subjects
  Arthralgia | 2 | 4
  Fatigue | 19 | 15
  Headache | 24 | 21
  Muscle aches | 15 | 17
  Shivering | 3 | 2
  Temperature ≥ 38.0°C | 1 | 0

3. Primary Outcome: Number of Subjects With Medically Attended Adverse Events (MAEs).
Description: Medically-attended events (MAEs) refer to non-serious and serious events leading to an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits and hospitalization. Related MAE = MAE assessed by the investigator as related to the vaccination.
Time Frame: During the entire study period (Days 0-182)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 101 | 99
subjects | 4 | 7

4. Primary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs).
Description: NOCDs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: During the entire study period (Days 0-182)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 101 | 99
subjects | 0 | 0

5. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: Unsolicited AEs cover any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any unsolicited AE = any unsolicited AE regardless of intensity or relationship to vaccination.
Time Frame: During the 90-day (Days 0-89) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 101 | 99
subjects | 28 | 21

6. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE = any SAE regardless of intensity or relationship to vaccination.
Time Frame: During the entire study period (Days 0-182)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 101 | 99
subjects | 1 | 0

7. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies for 3 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 3 influenza strains assessed were A/Solomon Islands/3/2006 (H1N1), A/Wisconsin/67/2005 (H3N2) and B/Malaysia/2506/2004 (MALAY.)
Time Frame: At Day 21
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 100 | 98
titers
  H1N1 | 183.7 [136.1 to 248.0] | 501.4 [397.8 to 632.0]
  H3N2 | 333.5 [278.5 to 399.3] | 315.5 [261.1 to 381.2]
  MALAY. | 316.6 [255.4 to 392.5] | 326.8 [264.9 to 403.3]

8. Primary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI antibody titer ≥ 1:40, a level of HI antibody that has been viewed as correlating with protection against influenza. The 3 influenza strains assessed were A/Solomon Islands/3/2006 (H1N1), A/Wisconsin/67/2005 (H3N2) and B/Malaysia/2506/2004 (MALAY.)
Time Frame: At Day 21
Population: as for outcome 7
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 100 | 98
subjects
  H1N1 | 90 | 97
  H3N2 | 98 | 98
  MALAY. | 99 | 96

9. Primary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 influenza strains assessed were A/Solomon Islands/3/2006 (H1N1), A/Wisconsin/67/2005 (H3N2) and B/Malaysia/2506/2004 (MALAY.)
Time Frame: At Day 21
Population: as for outcome 7
Measure: Number; unit: subjects
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 100 | 98
subjects
  H1N1 | 72 | 79
  H3N2 | 68 | 66
  MALAY. | 74 | 67

10. Primary Outcome: Geometric Mean Fold-rise (GMFR) in 3 Strains of Influenza Disease.
Description: GMFR was defined as the geometric mean of the ratio of the post-vaccination inverse HI titer to the Day 0 inverse HI titer. The 3 influenza strains assessed were A/Solomon Islands/3/2006 (H1N1), A/Wisconsin/67/2005 (H3N2) and B/Malaysia/2506/2004 (MALAY.)
Time Frame: At Day 0 and Day 21
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | GSK 1388442A Group | Fluarix Group
Number analyzed (Participants) | 100 | 98
fold rise
  H1N1 | 10.9 [8.0 to 14.9] | 17.8 [12.8 to 24.7]
  H3N2 | 10.1 [7.4 to 13.9] | 7.5 [5.6 to 10.1]
  MALAY. | 12.3 [9.0 to 16.8] | 10.5 [7.7 to 14.3]

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (Days 0-182); Unsolicited AE(s): during the 90-day (Days 0-89) post-vaccination period; Solicited local/general symptoms: during the 7-day (Days 0-6) post-vaccination period.
Arm/Group | GSK 1388442A Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 1/101 | 0/99
Other Adverse Events (participants affected / at risk) | 64/101 | 63/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 1388442A Group (N=101) | Fluarix Group (N=99)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK 1388442A Group (N=101) | Fluarix Group (N=99)
Pain (General disorders) | 48 | 48
Fatigue (General disorders) | 19/100 | 15
Headache (General disorders) | 24/100 | 21
Muscle aches (General disorders) | 15/100 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.